CLINICAL TRIAL: NCT00647790
Title: PET Using Hormone Receptor Ligands in Breast Cancer
Brief Title: Positron Emission Tomography (PET) Using Hormone Receptor Ligands in Breast Cancer
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 05-088
Record Dates: First submitted 2008-03-28; First posted 2008-04-01 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Breast Cancer
Keywords: PET imaging; invasive breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum blood sample postimaging, Serum Estradiol (female only)

GROUPS / COHORTS (1):
- 1: Patients with a confirmed diagnosis of invasive breast cancer who are undergoing surgery.
  Interventions: Procedure: PET scan with injection of 5-8 mCi of 18FES

INTERVENTIONS:
Procedure: PET scan with injection of 5-8 mCi of 18FES — Following injection of the tracer 18FES, dynamic images will be obtained for 30 minutes over the chest area to include cardiac region and breasts. Following the first dynamic imaging for 30 minutes, whole body images (base of skull to pelvis) will be obtained at 5 minute/bed position. An additional, longer scan after 60 minutes will be obtained for the chest (1-2-FOV for 15 minutes each). Total time from injection to completion of imaging will be about 90 minutes.

SUMMARY:
The purpose of this study is to find a way to learn the hormone receptor status of a tumor before surgery is done. By testing for the hormone receptor proteins, doctors can find out if the breast cancer uses hormones to grow. This is important since the hormone receptor status of a tumor helps doctors decide if extra treatment like chemotherapy or pills are needed.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female patients
* Aged 18 or older at the time of breast cancer diagnosis
* Patients with invasive breast cancer at least 1 cm in size. Patients who have had a prior surgical excision are eligible provided there is a residual of at least a 1 cm area suspected on imaging studies.
* Histopathologic review at MSKCC confirming diagnosis of invasive breast cancer (ductal, lobular, or inflammatory breast cancer).
* Patients who are operative candidates. Patient will have surgery to include either mastectomy or lumpectomy. Radiologic assisted excisions such as needle localization are also eligible.
* Patients with bilateral breast cancer are eligible.
* Patients with metastatic cancer, provided they need surgical biopsy.
* Patients who are undergoing sentinel node mapping (day before or sameday mapping).
* Patient must sign informed consent.

Exclusion Criteria:

* Previous or concurrent malignancy (except basal and squamous skin cancer and stage 0 cervical cancer)
* Patients who are pregnant or nursing
* Patients unable to tolerate PET or PET/CT
* Patients with known active infection, autoimmune or inflammatory disease such as sarcoidosis, and rheumatoid arthritis.
* Patients with non invasive breast cancer such as DCIS.
* Patients who have received prior radiation therapy to the affected breast.
* Patients who have received prior chemotherapy, including neoadjuvant chemotherapy or hormonal therapy for breast cancer.
* Patients living in a residential care or correctional facility.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast Clinic
Sampling Method: Non-Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2006-11; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
To use estrogen-like ligands labeled with positron emitters to preoperatively evaluate the estrogen receptor (ER) status of breast cancer on PET imaging. | conclusion of the study

SECONDARY OUTCOMES:
To correlate ER positivity on PET ligand imaging, and conventional immunohistochemical pathologic analysis of ER positivity in surgical specimens. | conclusion of the study

CONTACTS AND LOCATIONS:
Overall Officials: Mary Gemignani, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org